CLINICAL TRIAL: NCT03246529
Title: A Phase III, Randomized, Placebo-Controlled, Multi-Centre Study Evaluating the Safety, Tolerability and Efficacy of Combination Treatment of BL-8040 and G-CSF as Compared to Placebo and G-CSF for the Mobilization of Hematopoietic Stem Cells for Autologous Transplantation in Subjects With Multiple Myeloma - The GENESIS Study
Brief Title: A Phase III, Safety, Tolerability and Efficacy of Combination Treatment of BL-8040 and Granulocyte Colony Stimulating Factor (G-CSF) as Compared to Placebo and G-CSF for the Mobilization of Hematopoietic Stem Cells for Autologous Transplantation in Subjects With Multiple Myeloma (MM)
Acronym: GENESIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BL-8040.SCM.301
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 4-fluorobenzoyl-TN-14003; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Subjects were randomized using a 2:1 ratio to receive G-CSF + BL-8040 or G-CSF + Placebo, respectively. Randomization will use permuted blocks stratifying subjects by US geographical region (NorthEast, SouthEast, MidWest, SouthWest and NorthWest), remission status (CR vs. PR), and baseline platelet count (< 200 × 10^9/L or ≥ 200 × 10^9/L).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BL-8040 1.25 mg/kg + G-CSF (Experimental): Double-blind placebo-controlled setting designed to assess the safety, tolerability and efficacy of G-CSF + BL-8040 as compared to G-CSF + Placebo, for stem cell mobilization in MM.
  Interventions: Drug: BL-8040 1.25 mg/kg + G-CSF
- Placebo + G-CSF (Active Comparator): Double-blind placebo-controlled setting designed to assess the safety, tolerability and efficacy of G-CSF + BL-8040 as compared to G-CSF + Placebo, for stem cell mobilization in MM.
  Interventions: Drug: Placebo +G-CSF

INTERVENTIONS:
Drug: BL-8040 1.25 mg/kg + G-CSF — Up to 2 subcutaneous (SC) injections of BL-8040 are anticipated during the study. Injections of G-CSF per standard of care
  Arms: BL-8040 1.25 mg/kg + G-CSF
Drug: Placebo +G-CSF — Up to 2 SC injections of Placebo are anticipated during the study. Injections of G-CSF per standard of care
  Arms: Placebo + G-CSF

SUMMARY:
A total of 122 subjects were randomized into the study and investigated in the double-blind placebo-controlled setting to assess the efficacy and safety of G-CSF + BL-8040 as compared to G-CSF + placebo.

DETAILED DESCRIPTION:
* Part 1: This lead-in period, designed to ascertain the dose of BL-8040, enrolled a total of 12 subjects to an open labeled treatment to assess the efficacy, safety, pharmacokinetic (PK) and pharmacodynamic (PD) parameters of treatment with G-CSF 10 µg/kg/day and BL-8040 1.25 mg/kg, per study protocol to goal collection of ≥ 6 × 10^6 CD34+ cells/kg.
* Part 2: Following the successful completion of Part 1, a total of 122 subjects were randomized into Part 2 of the study which employed a double-blind placebo-controlled setting to assess the efficacy and safety of G-CSF + BL-8040 as compared to G-CSF + placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Multiple Myeloma prior to enrolment and randomization.
2. At least 1 week (7 days) from last induction cycle of combination/multi-agent cyto-reductive chemotherapy (e.g., KRD [carfilzomib, lenalidomide, dexamethasone] or VRD (e.g., bortezomib, lenalidomide, dexamethasone) or last single agent chemotherapy (e.g., lenalidomide, pomalidomide, bortezomib, dexamethasone, etc.) prior to the first dose of G-CSF for mobilization.
3. Eligible for autologous hematopoietic stem cell transplantation according to the Investigator's discretion.
4. The subjects should be in first or second CR (including CR and SCR) or PR (including PR and VGPR).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Adequate organ function at screening as defined as below:

   1. Hematology:

      * White blood cell counts more than 2.5 x 10^9/L
      * Absolute neutrophil count more than 1.5 x 10^9/L
   2. Platelet count more than 100 x10^9/L Renal Function:

      • Glomerular Filtration Rate (GFR) value of ≥15 mL/min/1.732 calculated by Modification of Diet in Renal Disease (MDRD) equation
   3. Hepatic function:

      * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x ULN
      * Total Bilirubin ≤ 2.0 x Upper Limit Normal (ULN) unless the subject has Gilbert disease
   4. Coagulation test:

      * International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 x ULN unless subject is receiving anticoagulant therapy, as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants
      * Activated Partial Thromboplastin Time (aPTT): ≤1.5 x ULN unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
7. Male subjects must agree to use an adequate method of contraception starting with the first day of G-CSF administration through 30 days after the last dose of study drug.
8. Patients must have a signed study informed consent prior to entering the study.

Exclusion Criteria:

1. Previous history of autologous or allogeneic-Hematopoietic Cell Transplantation (HCT).
2. Failed previous Hematopoietic Stem Cell (HSC) collections or collection attempts.
3. Taken any of the listed below concomitant medications, growth factors or stimulating agents within the designated washout period:

   1. Dexamethasone: 7 days;
   2. Thalidomide: 7 days;
   3. Lenalidomide: 7 days;
   4. Pomalidomide: 7 days;
   5. Bortezomib: 7 days;
   6. Carfilzomib: 7 days;
   7. G-CSF: 14 days;
   8. Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) or Neulasta®: 21 days;
   9. Erythropoietin or erythrocyte stimulating agents: 30 days;
   10. Eltrombopag, romiplostim or platelet stimulating agents: 30 days;
   11. Carmustine (BCNU): 42 days/6 weeks;
   12. Daratumumab: 28 days;
   13. Ixazomib: 7 days.
4. Received >6 cycles lifetime exposure to thalidomide or lenalidomide.
5. Received >8 cycles of alkylating agent combinations.
6. Received >6 cycles of melphalan.
7. Received prior treatment with radioimmunotherapy (e.g., radionuclides, holmium).
8. Received prior treatment with venetoclax.
9. Plans to receive maintenance treatment within 60 days post-engraftment (e.g., lenalidomide, bortezomib, pomalidomide, thalidomide, carfilzomib, etc.)
10. Has received a live vaccine within 30 days of the planned start of G-CSF administration. Seasonal flu vaccines that do not contain live virus are permitted.
11. Known active central nervous system (CNS) metastases or carcinomatous meningitis.
12. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to BL-8040, G-CSF, or other agents used in the study.
13. Has an active infection requiring systemic therapy or uncontrolled infection.
14. Has a known additional malignancy that is progressing or requires active treatment.
15. Has an underlying medical condition that would preclude study participation.
16. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
17. O2 saturation < 92% (on room air).
18. Personal history or family history of Long QT Syndrome or Torsade de Pointes.
19. History of unexplained syncope, syncope from an uncorrected cardiac etiology, or family history of sudden cardiac death.
20. Myocardial infarction, coronary artery bypass grafting (CABG), coronary or cerebral artery stenting and /or angioplasty, stroke, cardiac surgery, or hospitalization for congestive heart failure within 3 months or greater than Angina Pectoris Class >2 or New York Heart Association (NYHA) Heart Failure >2.
21. ECG in screening showing QTcF > 470 msec, and/or PR > 280 msec,.
22. Mobitz II 2nd degree Atrioventricular (AV) Block, 2:1 AV Block, High Grade AV Block, or Complete Heart Block, unless the patient has an implanted pacemaker or implantable cardiac defibrillator (ICD) with backup pacing capabilities.
23. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
25. Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 30 days after the last dose of study drug.
26. Has a known history of HIV (HIV 1/2 antibodies)
27. Has known active Hepatitis B (e.g., Hepatitis B Surface Antigen [HBsAg] reactive) or Hepatitis C (e.g., Hepatitis C Virus [HCV] RNA [qualitative] is detected).
28. Untreated or unsuccessfully treated Hepatitis B or C.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2029-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John DiPersio, MD, Principal Investigator — Washington University School of Medicine; Crees Zachary, MD, Principal Investigator — Washington University School of Medicine
Locations (18):
- United States (10):
  - UCLA Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - The Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston Texas, Texas
  - Huntsman Cancer Institute in University of Utah, Salt Lake City, Utah
- University of Koln, Cologne, Koln, Germany
- Hungary (2):
  - Central Hospital of Southern Pest National Institute of Hematology and Infectious Diseases, Budapest
  - University of Debrecen, Debrecen
- Italy (2):
  - Div. Clinicizzata di Ematologia - Policlinico Vittorio Emanuele, Catania
  - Presidio Ospedaliero Morelli Viale Europa, Reggio Calabria
- Spain (3):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital University Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crees ZD, Rettig MP, Jayasinghe RG, Stockerl-Goldstein K, Larson SM, Arpad I, Milone GA, Martino M, Stiff P, Sborov D, Pereira D, Micallef I, Moreno-Jimenez G, Mikala G, Coronel MLP, Holtick U, Hiemenz J, Qazilbash MH, Hardy N, Latif T, Garcia-Cadenas I, Vainstein-Haras A, Sorani E, Gliko-Kabir I, Goldstein I, Ickowicz D, Shemesh-Darvish L, Kadosh S, Gao F, Schroeder MA, Vij R, DiPersio JF. Motixafortide and G-CSF to mobilize hematopoietic stem cells for autologous transplantation in multiple myeloma: a randomized phase 3 trial. Nat Med. 2023 Apr;29(4):869-879. doi: 10.1038/s41591-023-02273-z. Epub 2023 Apr 17. PMID 37069359
- [Derived] Crees ZD, Stockerl-Goldstein K, Vainstein A, Chen H, DiPersio JF. GENESIS: Phase III trial evaluating BL-8040 + G-CSF to mobilize hematopoietic cells for autologous transplant in myeloma. Future Oncol. 2019 Nov;15(31):3555-3563. doi: 10.2217/fon-2019-0380. Epub 2019 Sep 9. PMID 31495201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 180 subjects signed the Informed Consent Form (ICF) and screened to the study. A total of 136 subjects received at least one dose of G-CSF. A total of 134 subjects were treated with G-CSF and with BL-8040 or Placebo.
Groups:
- BL-8040 + G-CSF Part 1: Part 1 (lead-in) period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- BL-8040 + G-CSF Part 2: Part 2: randomized, double-blinded, placebo controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- Placebo + G-CSF Part 2: Part 2: randomized, double-blinded, placebo controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. Placebo s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
Period: Core Study (until 100 d post-transplant)
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Started | 12 | 80 | 42
Post Transplantation Analysis Set | 12 | 77 | 37
Completed | 12 | 74 | 34
Not Completed | 0 | 6 | 8
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Other Reasons | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 4
Period: Follow-up period at 1 year FU Completion
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Started | 12 | 73 (One (1) subject early terminated the study following the core study period and before the follow up (FU)) | 34
Completed (Long Term FU is ongoing. Numbers are of the subject ongoing in the study.) | 9 | 66 | 32
Not Completed | 3 | 7 | 2
Not completed — Disease progression | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part 1: Full analysis set - all enrolled subjects. Part 2: ITT analysis set: all randomized subjects. According to the treatment group to which they were originally randomized.
Groups:
- Placebo + G-CSF Part 2: Part 2: randomized, double-blinded, placebo controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. Placebo s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- Total: Total of all reporting groups
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2 | Total
Number analyzed (Participants) | 12 | 80 | 42 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (4.8) | 60.4 (9.4) | 59.2 (9.6) | 60.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 25 | 18 | 48
  Male | 7 | 55 | 24 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2 | 8 | 2 | 12
  Caucasian | 9 | 65 | 40 | 114
  Not reported | 1 | 0 | 0 | 1
  African | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Hispanic origin | 0 | 1 | 0 | 1
  Unknown | 0 | 2 | 0 | 2
  Not Specified | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 0 | 10 | 6 | 16
  United States | 12 | 52 | 26 | 90
  Italy | 0 | 9 | 8 | 17
  Germany | 0 | 3 | 0 | 3
  Spain | 0 | 6 | 2 | 8
Treatment Indicated for Multiple Myeloma Before Study Initiation [Count of Participants; unit: Participants] — Treatment Indicated for Multiple Myeloma Before Study Initiation
  Participants
    Bortezomib | 7 | 54 | 28 | 89
    Cisplatin | 0 | 0 | 1 | 1
    Cyclophosphamide | 0 | 5 | 4 | 9
    Daratumumab 0 - 1 2.4% | 0 | 0 | 1 | 1
    Doxorubicin | 0 | 0 | 1 | 1
    Etoposide | 0 | 0 | 1 | 1
    Ixazomib | 0 | 1 | 0 | 1
    Kyprolis | 6 | 2 | 1 | 9
    Lenalidomide | 12 | 57 | 28 | 97
    Melphalan | 0 | 0 | 1 | 1
    Pomalidomide | 1 | 0 | 1 | 2
    Thalidomide | 0 | 18 | 12 | 30
IMWG Classification at Screening [Count of Participants; unit: Participants] — Response criteria for the purposes of the study was defined in accordance with the International Myeloma Working Group (IMWG) Uniform Response Criteria.
  Participants
    PR (Partial Response) | 0 | 31 | 10 | 41
    VGPR (Very Good Partial Response) | 9 | 33 | 23 | 65
    CR (Complete Response) | 2 | 12 | 7 | 21
    sCR (Stringent Complete Response) | 1 | 4 | 2 | 7
Months from MM Diagnosis to Study Consent [Mean (Standard Deviation); unit: months] | 4.6 (0.9) | 6.5 (11.1) | 6.4 (6.9) | 6.3 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Mobilizing ≥6 × 10^6 CD34+ Cells/kg With up to 2 Apheresis Sessions
Description: Percentage of subjects mobilizing ≥6 × 10^6 CD34+ cells/kg with up to 2 apheresis sessions in preparation for autologous hematopoetic cell transplantation (auto-HCT) after treatment with G-CSF + single administration of BL-8040/placebo.
  Based on central laboratory data.
Time Frame: From first day of study treatment (G-CSF) until day of second apheresis which was planned to occur on Day 6
Population: Full Analysis Set (FAS) for Part 1 (Part 1 of the study assessed the mobilization using local lab only), Intention-to-Treat (ITT) for Part 2
Measure: Number; unit: Percentage of responders
Groups:
- BL-8040 + G-CSF Part 1: Part 1 (lead-in) period. G-CSF given one time daily s.c. for 5-8 days (Days 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- BL-8040 + G-CSF Part 2: Part 2: randomized, double-blinded, placebo-controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- Placebo + G-CSF Part 2: Part 2: randomized, double-blinded, placebo-controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. Placebo s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 12 | 80 | 42
Percentage of responders
  Central Lab: number analyzed (Participants) | 0 | 80 | 42
  Central Lab |  | 70.0 | 14.3
  Local Lab | 91.7 | 92.5 | 26.2
Statistical Analysis 1: Comparison: BL-8040 + G-CSF Part 2 vs Placebo + G-CSF Part 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel (CMH) test (by response status and baseline platelet count),

2. Secondary Outcome: Percentage of Subjects Mobilizing ≥2 × 10^6 CD34+ Cells/kg in 1 Apheresis Session
Description: Percentage of subjects mobilizing ≥2 × 10^6 CD34+ cells/kg in 1 apheresis session after treatment with G-CSF + single administration of BL-8040/ placebo.
Time Frame: From first day of study treatment (G-CSF) until day of first apheresis which was planned to occur on Day 5
Population: FAS for Part 1 (Part 1 of the study assessed the mobilization using local lab only), ITT for Part 2
Measure: Number; unit: Percentage of responders
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 12 | 80 | 42
Percentage of responders
  Central Lab: number analyzed (Participants) | 0 | 80 | 42
  Central Lab |  | 87.5 | 47.6
  Local Lab | 100 | 96.3 | 64.3
Statistical Analysis 1: Comparison: BL-8040 + G-CSF Part 2 vs Placebo + G-CSF Part 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Subjects Mobilizing ≥6 × 10^6 CD34+ Cells/kg in 1 Apheresis Session
Description: Percentage of subjects mobilizing ≥6 × 10^6 CD34+ cells/kg in 1 apheresis session after treatment with G-CSF + single administration of BL-8040/ placebo.
Time Frame: From first day of study treatment (G-CSF) until day of first apheresis which was planned to occur on Day 5
Population: FAS for Part 1 (Part 1 of the study assessed the mobilization using local lab only), ITT for Part 2
Measure: Number; unit: Percentage of responders
Groups:
- BL-8040 + G-CSF Part 2: Part 2: randomized, double-blinded, placebo-controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4.
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 12 | 80 | 42
Percentage of responders
  Central Lab: number analyzed (Participants) | 0 | 80 | 42
  Central Lab |  | 67.5 | 4.8
  Local Lab | 75 | 88.8 | 9.5
Statistical Analysis 1: Comparison: BL-8040 + G-CSF Part 2 vs Placebo + G-CSF Part 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Time to Neutrophil Engraftment, After Auto-HCT
Description: Time to neutrophil engraftment after auto-HCT, where engraftment was defined as absolute neutrophil count (ANC) ≥0.5 × 10^9/L for 3 days or ≥1.0 × 10^9/L for 1 day following the conditioning regimen associated nadir.
Time Frame: End of engraftment period, which was defined as 29 days post transplantation
Population: Post Transplantation analysis set (all subjects treated, with at least 1 apheresis session, and who underwent transplantation)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 12 | 77 | 37
Days | 12 [11 to 12] | 12 [11 to 12] | 12 [11 to 12]

5. Secondary Outcome: Time to Platelet Engraftment, After Auto-HCT
Description: Time to platelet engraftment, after auto-HCT, where engraftment was defined as the first of 3 consecutive measurements of platelet count ≥20 × 10^9/L without platelet transfusion support for 7 days following the conditioning regimen associated nadir.
Time Frame: End of engraftment period, which was defined as 29 days post transplantation
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Point estimate (days)
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 12 | 77 | 37
Point estimate (days) | 17 [15.0 to 20.0] | 18 [17 to 19] | 17 [17 to 18]

6. Secondary Outcome: Subjects With Graft Durability at 100 Days Post Transplant/ Early Termination
Description: Subjects achieving graft durability were defined as meeting the following 2 criteria:
  * Platelet count ≥50 × 10^9/L without transfusion for at least 2 weeks.
  * Hemoglobin level ≥10 g/dL with no erythropoietin support or transfusions for at least 1 month.
  This analysis was performed in part 2 of the study only.
Time Frame: Day 100 Post-Transplantation (± 7 days)
Population: Post Transplantation analysis set (all randomized subjects treated, with at least 1 apheresis session, and who underwent transplantation).
  Graft durability was not assessed during Part 1 of the study.
Measure: Number; unit: Percentage of responders
Arm/Group | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 77 | 37
Percentage of responders | 92.2 | 91.9

7. Secondary Outcome: Graft Durability at 6 Months Post Transplantation
Description: Comparability of the graft durability between the BL-8040 + G-CSF arm and the placebo + G-CSF arm at 6 months post transplantation
Time Frame: 6 Months Post Transplantation
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Groups:
- BL-8040 + G-CSF Part 2; Placebo + G-CSF Part 2: Part 2: Randomized, double-blind, placebo-controlled period
Arm/Group | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 77 | 37
Percentage of responders | 80.5 | 83.8

8. Secondary Outcome: Graft Durability at 9 Months Post Transplantation
Description: Comparability of the graft durability between the BL-8040 + G-CSF arm and the placebo + G-CSF arm at 9 months post transplantation
Time Frame: 9 Months Post Transplantation
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 77 | 37
Percentage of responders | 83.1 | 81.1

9. Secondary Outcome: Graft Durability at 12 Months Post Transplantation
Description: Comparability of the graft durability between the BL-8040 + G-CSF arm and the placebo + G-CSF arm at 12 months post transplantation
Time Frame: 12 Month Post Transplantation
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | BL-8040 + G-CSF Part 2 | Placebo + G-CSF Part 2
Number analyzed (Participants) | 77 | 37
Percentage of responders | 81.8 | 81.1

10. Other Pre Specified Outcome: Overall Survival Until September 2028
Description: Comparability between the effect of BL-8040 + G-CSF and placebo + G-CSF on Overall Survival until September 2028
Time Frame: End of Study
Reporting Status: Not Posted, anticipated posting 2029-06

11. Other Pre Specified Outcome: Relapse Free Survival Until September 2028
Description: Comparability between the effect of BL-8040 + G-CSF and placebo + G-CSF on Relapse Free Survival until September 2028
Time Frame: End Of Study
Reporting Status: Not Posted, anticipated posting 2029-06

12. Other Pre Specified Outcome: Annualized Relapse Rate Until September 2028
Description: Comparability between the effect of BL-8040 + G-CSF and placebo + G-CSF on Annualized Relapse Rate until September 2028
Time Frame: End of Study
Reporting Status: Not Posted, anticipated posting 2029-06

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected after subjects signed the ICF and up to 30 days from the last dose of study therapy (G-CSF+BL-8040/Placebo).
Description: All AEs were collected after subjects signed the ICF and up to 30 days from the last dose of study therapy (G-CSF+BL-8040/Placebo). AE were followed by the investigators until their satisfactory resolution or stabilization. AE were recorded and graded according to the latest version of the NCI-CTCAE.
  All-cause mortality was reported across the entire study duration, including the 5 years follow-up phase.
Groups:
- BL-8040 + G-CSF (Part 2): Part 2: randomized, double-blinded, placebo-controlled period. G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. BL-8040 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
- Placebo + G-CSF (Part 2): Part 2 (randomized, double-blinded, placebo-controlled period). G-CSF given one time daily s.c. for 5-8 days (Day 1 up to 8) at doses of approximately 10 µg/kg/day but not more than 15 µg/kg/day. Placebo 1.25 mg/kg s.c. on Day 4 (and Day 6, if needed).
  First apheresis on Day 5 with up to 3 additional procedures possible until Day 8, as needed.
Arm/Group | BL-8040 + G-CSF Part 1 | BL-8040 + G-CSF (Part 2) | Placebo + G-CSF (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/12 | 2/80 | 1/42
Serious Adverse Events (participants affected / at risk) | 1/12 | 7/80 | 0/42
Other Adverse Events (participants affected / at risk) | 12/12 | 77/80 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BL-8040 + G-CSF Part 1 (N=12) | BL-8040 + G-CSF (Part 2) (N=80) | Placebo + G-CSF (Part 2) (N=42)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BL-8040 + G-CSF Part 1 (N=12) | BL-8040 + G-CSF (Part 2) (N=80) | Placebo + G-CSF (Part 2) (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 14 (17) | 6 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 14 (15) | 13 (18)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Auricular swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 9 (9) | 6 (6)
Chest pain (General disorders) | 1 (1) | 2 (3) | 4 (5)
Injection site erythema (General disorders) | 3 (3) | 22 (22) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 9 (14) | 40 (47) | 2 (3)
Injection site pruritus (General disorders) | 5 (6) | 17 (17) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 5 (5) | 0 (0)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 3 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 11 (11) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 6 (6) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 11 (11) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (5)
Paraesthesia (Nervous system disorders) | 1 (1) | 8 (11) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 5 (6) | 3 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (15) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 26 (28) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (10) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 0 (0)
Flushing (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restrictions are as per the signed agreement with each PI and institution.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03246529/Prot_SAP_000.pdf